CLINICAL TRIAL: NCT04328389
Title: Periodontal Management in Hypertensive Patients
Brief Title: Periodontal Management in Hypertensive Patients (PERIOTENSION Trial I)
Acronym: PERIOTENSION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of L'Aquila (Other)
Responsible Party: Principal Investigator, Davide Pietropaoli, junior researcher, University of L'Aquila
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AQ2020
Record Dates: First submitted 2020-03-27; First posted 2020-03-31 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Periodontal Diseases; Gingivitis; Hypertension
MeSH Terms: conditions — Periodontal Diseases; Gingivitis; Hypertension

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Comparator: electric toothbrush (Placebo Comparator): Participats will be instructed to used electric toothbrush for home supragingival plaque removal
  Interventions: Behavioral: electric toothbrush
- Professional oral hygiene (Experimental): Full-Mouth professional oral hygiene consisting in scaling and root planing, four quadrants in one session.
  Interventions: Procedure: Professional oral hygiene

INTERVENTIONS:
Behavioral: electric toothbrush — Participants will be instructed to use their electric toothbrushes twice a day for controlling oral plaque
  Arms: Placebo Comparator: electric toothbrush
Procedure: Professional oral hygiene — Professional oral hygiene using ultrosound scaling and root planing
  Arms: Professional oral hygiene

SUMMARY:
Treated hypertensive patients with any form of periodontal diseases will be randomized to either supragingival dental plaque removal using electric toothbrushes at home or intensive professional oral hygiene treatment and the effects on blood pressure will be identified.

ELIGIBILITY:
Inclusion Criteria:

* Treated hypertension
* Have at least 20 natural teeth
* Presence of any form of periodontal diseases according to guidelines
* Absence of other significant oral infections.

Exclusion Criteria:

* Secondary hypertension (known plasma renin screening, abdominal ultrasound with doppler and other investigations)
* Individual is pregnant or nursing
* Primary pulmonary hypertension
* Professional oral hygine within past 6 months
* Flu, rhinitis, sinusitis etc. within past 4 weeks
* Use of antibiotics within past 4 weeks
* Hospitalization for any reason within the past 3 months
* Allergic disorders; History of chronic infectious disease,
* Chronic hepatitis B or C infection
* Chronic Obstructive Pulmonary Disease (COPD), tuberculosis
* Other known chronic inflammatory or autoimmune condition such as lupus or rheumatoid arthritis, ulcerative colitis or Crohn's disease
* Use of systemic or local steroids or immunosuppressive agents within 6 months of the inclusion.
* History of alcohol abuse or unwillingness to limit alcohol consumption to less than 4 drinks per week

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Systolic and Diastolic Blood Pressure Change | 1 week
  Ambulatory Blood Pressure Monitoring

SECONDARY OUTCOMES:
Systolic and Diastolic Blood Pressure Change | 1 week
  Unattented Blood Pressure Measurement

OTHER OUTCOMES:
Periodontal Health Score - Bleeding on probing (BoP) | 1 week
Periodontal Health Score - Periodontal Probing Depth (PPD) | 1 week
Periodontal Health Score - Clinical Attachment Loss (CAL) | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Rita Del Pinto, MD, PhD, Principal Investigator — University of L'Aquila Unit of Internal Medicine and Nephrology - Center for Hypertension; Davide Pietropaoli, DDS, PhD, Principal Investigator — University of L'Aquila - Unit of Oral Diseases

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pietropaoli D, Del Pinto R, Ferri C, Wright JT Jr, Giannoni M, Ortu E, Monaco A. Poor Oral Health and Blood Pressure Control Among US Hypertensive Adults. Hypertension. 2018 Dec;72(6):1365-1373. doi: 10.1161/HYPERTENSIONAHA.118.11528. PMID 30540406
- [Background] Pietropaoli D, Del Pinto R, Ferri C, Ortu E, Monaco A. Definition of hypertension-associated oral pathogens in NHANES. J Periodontol. 2019 Aug;90(8):866-876. doi: 10.1002/JPER.19-0046. Epub 2019 May 29. PMID 31090063
- [Background] Pietropaoli D, Del Pinto R, Ferri C, Marzo G, Giannoni M, Ortu E, Monaco A. Association between periodontal inflammation and hypertension using periodontal inflamed surface area and bleeding on probing. J Clin Periodontol. 2020 Feb;47(2):160-172. doi: 10.1111/jcpe.13216. Epub 2019 Nov 26. PMID 31680283